CLINICAL TRIAL: NCT04830189
Title: Comparison of the Effectiveness of Two Different Types of Slings in Shoulder Subluxation
Brief Title: The Effectiveness of Two Different Types of Shoulder Slings in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstPMRTRH-BMR20
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Hemiplegia; Rehabilitation
Keywords: Stroke; subluxation; shoulder; slings
MeSH Terms: conditions — Hemiplegia; Stroke; Joint Dislocations

STUDY DESIGN:
Intervention Model Description: Patients were assigned to two groups, shoulder supported slings (group 1, n = 20) and forearm supported slings (group 2, n = 20), by an investigator who was blinded to the study via randomization created by a computer software. Evaluation of the detailed physical examination results, evaluation of demographic features such as age, gender, and etiology as well as evaluation of treatment results were performed by the physiatrist who was blind to randomization.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shoulder slings (Experimental): Patients were used shoulder sling in addition to conservative treatment.
  Interventions: Device: shoulder sling
- forearm sling (Active Comparator): Patients were used forearm sling in addition to conservative treatment.
  Interventions: Device: forearm sling

INTERVENTIONS:
Device: shoulder sling — Patients were used shoulder slings
  Arms: shoulder slings
Device: forearm sling — Patients were used forearm slings
  Arms: forearm sling

SUMMARY:
The aim of this study is to investigate the effectiveness of shoulder slings on pain, motor function, daily life and balance in acute hemiplegic patients and to investigate whether different types of slings are superior to each other.

DETAILED DESCRIPTION:
Thirty-two patients with hemiplegic shoulder subluxation due to acute stroke were divided into two groups: shoulder supported slings and forearm supported slings. Hemiplegia rehabilitation passive and active-assistive range of motion, stretching, and neurophysiologic exercises were performed for all patients per day for 8 weeks.Pain assessment was performed with Visual Analog Scale, sensorimotor evaluation was performed with Fugl Meyer Assessment of Motor Function,daily life activities were assessed with Barthel Index, and balance was evaluated with Berg Balance Scale.

ELIGIBILITY:
Inclusion Criteria:

* Acute patients who were independent and ambulatory prior to stroke and had their first stroke attack (<3 months)
* Mini-mental Status Test (MMST) score ≥ 24,
* Developing hemiplegia after stroke, standing independently for at least 2 minutes,
* Lower limb being in stage 4-5 according to the Brunnstrom Approach (for ambulation and standard balance)
* Upper limb being in stage 1-2 according to the Brunnstrom Approach
* Spasticity 0-1+ according to Modified Ashworth scale

Exclusion Criteria:

* Has a neurological history other than the diagnosis of hemiplegia (Parkinson's etc.)
* Having used shoulder slings and orthosis.
* Having a disease that can affect balance (cranial, etc.)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from Baseline VAS score at 8 weeks
  Pain assessment was performed with Visual Analog Scale after 8-weeks after treatment. Using a ruler, the score is determined by measuring the distance (mm) on the 100-mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Fugl-Meyer Assessment of Motor Recovery after Stroke | Change from Baseline Fugl Meyer test score at 8 weeks
  Sensorimotor evaluation was performed with Fugl-Meyer Assessment of Motor Recovery after Stroke. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Barthel Index | Change from Baseline Barthel Index score at 8 weeks
  Daily life activities were assessed with Barthel Index. The minimum score is 0, which indicates complete dependency and, the maximum score is 100 indicates complete independence.
Berg Balance Scale (BBS) | Change from Baseline Berg Balance Scale score at 8 weeks
  Balance was evaluated with Berg Balance Scale. The minimum score is 0 and, the maximum score is 56. 0-20 on the BBS represents balance impairment; 21-40 on the BBS represents acceptable balance; 41-56 on the BBS represents good balance.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Aziz Yıldırım, Assoc prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalichman L, Ratmansky M. Underlying pathology and associated factors of hemiplegic shoulder pain. Am J Phys Med Rehabil. 2011 Sep;90(9):768-80. doi: 10.1097/PHM.0b013e318214e976. PMID 21430513
- [Result] Zorowitz RD. Recovery patterns of shoulder subluxation after stroke: a six-month follow-up study. Top Stroke Rehabil. 2001 Summer;8(2):1-9. doi: 10.1310/LADU-8LJY-KTQ0-L5DJ. PMID 14523741
- [Result] Brooke MM, de Lateur BJ, Diana-Rigby GC, Questad KA. Shoulder subluxation in hemiplegia: effects of three different supports. Arch Phys Med Rehabil. 1991 Jul;72(8):582-6. PMID 2059138
- [Result] Williams R, Taffs L, Minuk T. Evaluation of two support methods for the subluxated shoulder of hemiplegic patients. Phys Ther. 1988 Aug;68(8):1209-14. PMID 3399517
- [Result] Turner-Stokes L, Jackson D. Assessment of shoulder pain in hemiplegia: sensitivity of the ShoulderQ. Disabil Rehabil. 2006 Mar 30;28(6):389-95. doi: 10.1080/09638280500287692. PMID 16492635
- [Result] Nadler M, Pauls M. Shoulder orthoses for the prevention and reduction of hemiplegic shoulder pain and subluxation: systematic review. Clin Rehabil. 2017 Apr;31(4):444-453. doi: 10.1177/0269215516648753. Epub 2016 Jul 10. PMID 27184582
- [Result] Ada L, Foongchomcheay A, Canning C. Supportive devices for preventing and treating subluxation of the shoulder after stroke. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003863. doi: 10.1002/14651858.CD003863.pub2. PMID 15674917
- [Result] van Bladel A, Lambrecht G, Oostra KM, Vanderstraeten G, Cambier D. A randomized controlled trial on the immediate and long-term effects of arm slings on shoulder subluxation in stroke patients. Eur J Phys Rehabil Med. 2017 Jun;53(3):400-409. doi: 10.23736/S1973-9087.17.04368-4. Epub 2017 Jan 30. PMID 28145396